CLINICAL TRIAL: NCT07148219
Title: Embrace Your Power: A VR Journey to Overcoming Negative Emotions for Romanian Youth
Brief Title: EMBRACE YOUR POWER
Acronym: EYP-VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Collaborators: Remnant Dream SRL (Unknown)
Responsible Party: Principal Investigator, Cezar Giosan, Cezar Giosan, PhD, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09242025
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Bullying; Distress; Bullying Victimisation
Keywords: randomized controlled trial; bullying; virtual reality; distress
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial where participants are divided into 2 groups: the intervention group that has access to the virtual reality program for preventing bullying and the inactive control group that receives the intervention after the study ends.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): VR program for preventing and combating bullying
  Interventions: Behavioral: Embrace Your Power: A VR Journey to Overcome Negative Emotions
- Waitlist (No Intervention): The control group receives the intervention after the study ends.

INTERVENTIONS:
Behavioral: Embrace Your Power: A VR Journey to Overcome Negative Emotions — EYP-VR represents a virtual reality (VR) educational tool to combat bullying. Using Meta Quest 3 passthrough technology, the app combines real-world classroom elements with immersive virtual scenarios, enabling safe and interactive experiences that simulate bullying situations but that do not place students in the roles of victims or aggressors but heroes or protectors.
  The app guides participants through narrative episodes focused on building empathy, practicing assertiveness, and learning conflict resolution techniques. AI-driven characters dynamically respond to students' actions as they engage in puzzles, and sensory feedback (visual, auditory, and haptic) reinforces key socio-emotional learning outcomes.
  The program will take place in classrooms during instructional hours. Each session will end with a feedback phase so that the school counselor can manage any issues that interest them.
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of an educational tool, based on virtual reality (VR), for preventing and combating bullying and for improving the emotional well-being of pre-adolescent students.

Participants will be allocated to one of two conditions:

* (1) intervention group: Embrace your power intervention for combating bullying;
* (2) waitlist (inactive control): the control group receives intervention after the study ends.

The intervention group will be compared to the control group in terms of peer aggression and victimization (bullying behaviors) and emotional symptoms.

DETAILED DESCRIPTION:
This protocol outlines a cluster, parallel-group, exploratory, randomized controlled trial where participants are randomly allocated to one of the two groups: intervention or control.

* The main objective is to implement and assess the effectiveness of the program for combating bullying through virtual reality. The program aims to reduce victimization and bullying behaviors (physical, verbal, and relational aggression) by applying the APRI tool as a result of participating in VR scenarios that simulate these situations and to reduce emotional difficulties and behavioral problems, as well as increase prosocial behavior.
* The included classes will serve as the randomization units. Students aged between 10 and 14 years, (5th and 6th grades from middle schools) will participate in the study. The intervention will last 7 weeks, and the two groups will be assessed at (1) pre-intervention (baseline), (2) middle of the intervention (week 3 or 4), and (3) post-intervention. The data analysis will focus on improvement in outcomes between and within groups.

ELIGIBILITY:
Inclusion Criteria:

* Students 5th and 6th grade
* Students whose parents have given their consent and who have also agreed to participate in the program

Exclusion Criteria:

* Medical problems that have VR-based procedures as contraindicated because they can induce dizziness, seizures, nausea:

  1. epilepsy
  2. presence of seizures
  3. severe motion sickness- vestibular disorders
  4. significant vision problems that would interfere with the use of the headset
  5. severe migraines triggered by exposure to screens
* Neurodevelopmental disorders

  1. Autism spectrum disorder- level 3 of severity or sensory processing disorders
  2. ADHD, if hyperactivity would prevent the student from staying in the exercise for longer
* Points a) and b) do not represent automatic exclusion criteria, because depending on the judgment of the school counselor, the parent and the teacher, it is possible that a participant will be able to complete the program.
* Severe mental disorders: psychotic spectrum disorders, post-traumatic stress disorder, present suicidal ideation
* If children have an extremely low level of literacy perceived by the teacher and counselor, and this aspect would prevent them from participating in the program.
* Parallel participation in other bullying prevention programs.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Bullying behaviors | Pre-intervention (baseline), middle intervention, post-intervention (week 7)
  Bullying behaviors will be measured using the Adolescent Peer Relations Instrument (APRI) -C2. The instrument encompasses bullying victimization, perpetration, and bystander experiences. APRI represents a psychometric tool that measures teens' experiences with bullying and victimization through 36 items rated on a 6-point Likert scale (1= never, 6= every day).

SECONDARY OUTCOMES:
Emotional symptoms | Pre-intervention (baseline), middle intervention, post-intervention (week 7)
  Emotional distress will be assessed using the Emotional Symptoms subscale from the Strengths and Difficulties Questionnaire - SDQ (Romanian self-report). The instrument consists of 25 items, and 5 items are representative of emotional symptoms. Items are rated on a 3-point Likert scale where 1= untrue and 3= certainly true.

OTHER OUTCOMES:
Strengths and Difficulties | Pre-intervention (baseline), middle intervention, post-intervention (week 7)
  The other subscales from the Strengths and Difficulties Questionnaire (SDQ) will be used to measure conduct problems (5 items), hyperactivity/inattention (5 items), peer relationship problems (5 items) and prosocial behavior (5 items). Items are measured on a 3-point Likert scale where 1= untrue and 5= certainly true.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided